CLINICAL TRIAL: NCT01450111
Title: Single-site, Randomized, Double-blind, Placebo-controlled, Parallel-group, Single/Repeated Dose Trial to Evaluate the Pharmacokinetics and Safety/Tolerability of Lacosamide in 3 Dosages in Healthy Male Korean Subjects
Brief Title: To Evaluate the Pharmacokinetics and Safety/Tolerability of Lacosamide in 3 Dosages in Healthy Male Korean Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SP0952
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Epilepsy
Keywords: Lacosamide
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Lacosamide 50 mg group (Experimental): Lacosamide 50 mg tablet, once a day per os (po)
  Interventions: Drug: Lacosamide
- Placebo group matched with lacosamide 50 mg (Placebo Comparator): Placebo matched with lacosamide 50 mg tablet, po
  Interventions: Other: Placebo
- Lacosamide 100 mg group (Experimental): Lacosamide 100 mg tablet, po
  Interventions: Drug: Lacosamide
- Placebo group matched with lacosamide 100 mg (Placebo Comparator): Placebo matched with lacosamide 100 mg tablet, po
  Interventions: Other: Placebo
- Lacosamide 200 mg group (Experimental): Lacosamide 200 mg tablet, po
  Interventions: Drug: Lacosamide
- Placebo group matched with lacosamide 200 mg (Placebo Comparator): Placebo matched with lacosamide 200 mg tablet, po
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lacosamide — Lacosamide 50 mg, tablet, once in the morning on Day 1
  Other Names: Vimpat®
  Arms: Lacosamide 50 mg group
Drug: Lacosamide — Lacosamide 100 mg, tablet, once in the morning on Day 1 Lacosamide 100 mg, tablet, twice daily Day 5 to Day 8 and once in the morning on Day 9
  Other Names: Vimpat®
  Arms: Lacosamide 100 mg group
Drug: Lacosamide — Lacosamide 200 mg, tablet, once in the morning on Day 1 Lacosamide 200 mg, tablet, twice daily Day 5 to Day 8 and once in the morning on Day 9
  Other Names: Vimpat®
  Arms: Lacosamide 200 mg group
Other: Placebo — Placebo matched with Lacosamide 50 mg tablet once in the morning on day 1.
  Arms: Placebo group matched with lacosamide 50 mg
Other: Placebo — Placebo matched with Lacosamide 100 mg, tablet, once in the morning on Day 1 Placebo matched with Lacosamode 100 mg, tablet, twice daily Day 5 to Day 8 and once in the morning on Day 9
  Arms: Placebo group matched with lacosamide 100 mg
Other: Placebo — Placebo matched with Lacosamide 200 mg, tablet, once in the morning on Day 1 Placebo matched with Lacosamide 200 mg, tablet, twice daily Day 5 to Day 8 and once in the morning on Day 9
  Arms: Placebo group matched with lacosamide 200 mg

SUMMARY:
Primary objective of this trial was to investigate the pharmacokinetics of single dose and repeated dose applications of lacosamide in healthy male Korean subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy male and between 20 and 45 years of age (inclusive)
* Subject has no clinically relevant cardiovascular, renal, gastrointestinal, hepatic, metabolic, endocrine, neurological, or psychiatric abnormalities and is in general good health
* Subject is of normal body weight as determined by a body mass index (BMI) between 19 and 28 kgm^2
* Subject is Korean (both parents are of pure Korean ethnicity)

Exclusion Criteria:

* Subject has a history of or present psychiatric or neurological condition that, in the opinion of the Investigator, could jeopardize or would have compromised the subject's ability to participate in this trial
* Subject has a known or suspected drug hypersensitivity, in particular to the trial medication
* Subject consumes more than 40 g alcohol/day (amount corresponds to 1 L beer/day or 0.5 L wine/day or 6 glasses (à 2cL) liquor/day)
* Subject has donated blood or had a comparable blood loss (>400 mL) within the last 3 months prior to Eligibility Assessment (EA)
* Subject smokes more than 5 cigarettes per day or had done so within 6 months prior to EA.
* Subject consumes more than 600 mg caffeine/day (200 mL coffee contain approximately 100 mg caffeine, 200 mL black tea approximately 30 mg, and 200 mL cola approximately 20 mg)
* Subject has a diet which deviates notably from the "normal" amounts of protein, carbohydrate, and fat, as judged by the Investigator (eg, vegetarians or vegans)
* Subject has taken herbal medicine therapy within 2 weeks prior to the first dosing
* Subject has a clinically relevant allergy
* Subject is taking any concomitant medication currently or within 2 weeks prior to the first dosing (with the exception of acetaminophen which is allowed to be taken orally up to 1000 mg per dose up to 48 hours prior to commencement of dosing)
* Subject has positive tests for alcohol and/or drugs (urine test) at EA and at confinement
* Subject has a high risk behavior for the HIV
* Subject is tested to be positive for HIV antibodies (HIV Ab), hepatitis B surface antigen (HBs Ag), or hepatitis C virus antibody (HCV Ab)
* Subject has a history or present condition of hepatic disorders, eg, clinically relevant liver enzyme increase (alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [AP], and gamma-glutamyl transpeptidase [GGT])
* Subject has a transaminase (either ALT or AST) more than 2 times of the upper limit of normal range (ULN) at confinement
* Subject has clinically relevant out-of-range values for hematology including coagulation parameters, and clinical chemistry, serology or urinalysis parameters
* Subject has any clinically relevant abnormality in the physical examination or vital signs
* Subject has a pulse rate at rest less than 45 bpm or more than 100 bpm at EA
* Subject has a systolic blood pressure lower than 100 mmHg or higher than 160 mmHg or a diastolic blood pressure higher than 95 mmHg at EA
* Subject has clinically relevant findings in the ECG, such as second or third degree atrioventricular (AV) block or PR interval >220 ms, prolongation of the QRS duration to >110 ms, or a QTcB (Bazett corrected) interval over 450 ms or any other clinically relevant ECG finding at EA
* Subject performed heavy physical exertion 2 days before EA or before confinement
* Subject has a history or present condition of respiratory or cardiovascular disorders, eg, cardiac insufficiency, coronary heart disease, hypertension, arrhythmia, tachyarrhythmia, or status after myocardial infarction
* Subject has a history or present condition of malignancy
* Subject has a history or present condition of seizure disorder
* Subject has atrial fibrillation/flutter, ventricular tachyarrhythmia (eg, ventricular tachycardia, ventricular fibrillation, aborted cardiac arrest), symptomatic heart block at Eligibility Assessment Visit, or is diagnosed with Brugada syndrome (also known as Sudden Unexpected Death Syndrome)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of lacosamide at steady state (Cmax) during up to 9 days of administration | Pharmacokinetic samples were taken pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84 and 96 hours after the first administration (at Day 1 & Day 9) and immediately before all administrations (at Day 5~8)
Time of maximum plasma concentration (Tmax) during up to 9 days of administration | Pharmacokinetic samples were taken pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84 and 96 hours after the first administration (at Day 1 & Day 9) and immediately before all administrations (at Day 5~8)
Area under the plasma concentration curve (AUC) during up to 9 days of administration | Pharmacokinetic samples were taken pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84 and 96 hours after the first administration (at Day 1 & Day 9) and immediately before all administrations (at Day 5~8)
The fraction of drug excreted unchanged in urine (Fe) during up to 9 days of administration | Urine samples were collected 0 - 4 hr, 4 - 8 hr, 8 - 12 hr, 12 - 24 hr, 24 - 48 hr, 48 - 72 hr, 72 - 96 hr after administration at Day 1 and Day 9

SECONDARY OUTCOMES:
Apparent clearance (CL/F) | Pharmacokinetic samples were taken pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84 and 96 hours after the first administration (at Day 1 & Day 9) and immediately before all administrations (at Day 5~8)
Apparent volume of distribution (V/F) | Pharmacokinetic samples were taken pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84 and 96 hours after the first administration (at Day 1 & Day 9) and immediately before all administrations (at Day 5~8)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)